CLINICAL TRIAL: NCT02245165
Title: Nitric Oxide Control of the Migrating Motor Complex in Man: L-NMMA Effects in Relation to Muscarinic and Serotonergic Receptor Blockade
Brief Title: Nitric Oxide Control of Migrating Motor Complex: L-NMMA Effects in Relation to Receptor Blockades
Acronym: LNMMA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Bengt Ihre Foundation (Other); The Swedish Society of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LNMMA-UU-02; LNMMA-UU-02 (Other Grant/Funding Number: Uppsala Univ, Bengt Ihre Fund, Swedish Soc of Medicine)
Record Dates: First submitted 2014-05-05; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Gastrointestinal Motility Disorder; Disturbance of Salivary Secretion
Keywords: Nitric oxide; Nitric oxide synthase; Gastrointestinal motility; Gut peptide hormones
MeSH Terms: interventions — omega-N-Methylarginine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitric oxide synthase (NOS) inhibition (Experimental): After a control period of 4 hours, intervention with L-NMMA (10 mg/kg IV) is done and recording continued for 4 hours.
  Interventions: Biological: L-Nitro-Monomethyl-Arginine (LNMMA) 10 mg/kg IV
- Saline (Sham Comparator): After a control period of 4 hours, intervention with saline is done and recording continued for 4 hours.
  Interventions: Biological: saline

INTERVENTIONS:
Biological: L-Nitro-Monomethyl-Arginine (LNMMA) 10 mg/kg IV
  Other Names: L-NMMA
  Arms: Nitric oxide synthase (NOS) inhibition
Biological: saline
  Arms: Saline

SUMMARY:
The aim is to elucidate how NO works in conjunction with other neurotransmitters to regulate the migrating motility complex (MMC). Twenty-two healthy volunteers should undergo water-perfused antroduodenojejunal manometry during a control period of 4 h, followed by another 4h after a bolus injection of either saline or the NO synthase inhibitor NG-monomethyl-L-arginine (L-NMMA, 10 mg/kg intravenously) with or without atropine (1 mg) or ondansetron (8 mg). Effects on the MMC pattern are determined. Exhaled and rectal NO is monitored throughout the experiments. Effects of L-NMMA on the MMC pattern are analyzed against a background of atropine or ondansetron. Blood samples are drawn for analysis of simultaneous peptide hormone release into the bloodstream. Peptide hormone release will be correlated to the respective motility pattern elicited by LNMMA.

DETAILED DESCRIPTION:
Dysregulation of the cyclic motility pattern controlling propulsion during fasting, the migrating motor complex (MMC), can result in small intestinal bacterial overgrowth and symptoms of intestinal obstruction. Nitric oxide (NO) acts as an inhibitory neurotransmitter by relaxation of smooth muscle cells. Little is known on how NO works in conjunction with other neurotransmitters to regulate the MMC.

Methods: Twenty-two healthy volunteers (22-38 years) should undergo antroduodenojejunal manometry recordings for 8h, 4h of which as a control period with basal motility recording and 4h after a bolus injection of either saline or the NO synthase inhibitor NG-monomethyl-L-arginine (L-NMMA, 10 mg/kg intravenously) with or without atropine (1 mg) or ondansetron (8 mg). The effects of L-NMMA on the MMC pattern are to be determined. Exhaled and rectal NO was monitored throughout the experiments as a means to secure efficient NO synthase inhibition.

Expected results: L-NMMA is expected to increase the intestinal motor activity, either as a direct effect on the small muscle cells, or through the release of some motility-stimulating gut peptide hormone (motility, ghrelin, somatostatin).

Expected conclusions: A NO donor, such as nitrite or nitrate which is converted to NO in an acidic milieu in the stomach may act as an inhibitor of motility. Thus, swallowed nitrite and nitrate from the saliva may contribute to the regulation of gastric emptying and gastrointestinal motility.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers 18-50 years of age

Exclusion Criteria:

* Age < 18, or > 50 years
* Any disease
* Any medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Effect on phases I-III of the migrating motor complex | 1 year
  NO is considered to be of importance for gastrointestinal motility. The MMC is measured as a biomarker of regulatory functions of gastrointestinal motility. Inhibition of the elaboration of NO by use of LNMMA is used to draw conclusions about the importance of NO for regulation of gastrointestinal motility.

SECONDARY OUTCOMES:
Reduced exhaled NO after administration of NO synthase inhibitor LNMMA | 1 year
  After administration of a Nitric oxide synthase (NOS) inhibitor exhaled NO is used as a marker of reduced NOS activity.

CONTACTS AND LOCATIONS:
Overall Officials: Per M Hellstrom, MD, prof, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Uppsala County, Sweden